CLINICAL TRIAL: NCT05901181
Title: The Effect of Laughter Yoga on Self-Care, Quality of Life and Stress Level in Menopause: A Randomized Controlled Study
Brief Title: The Effect of Laughter Yoga on Self-Care, Quality of Life and Stress Level in Menopause
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Dilek Karaoğlan, SENIOR INSTRUCTOR, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ETK00-2023-0059
Record Dates: First submitted 2023-05-22; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Laughter; Menopause; Stress; Self
Keywords: Laughter Yoga; Menopause; Stress; Self Care
MeSH Terms: conditions — Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: study design Applications of women will be received by making announcements of the research and laughter yoga trainings through posters hung in the center of the district to menopausal women in the 45-60 age group in the district. After the applications, menopausal women who meet the research criteria and volunteer to participate in the research will be randomly assigned to the intervention and control groups by drawing lots to determine which group they will be in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Yoga Group (Experimental): When we look at the literature, the Laughter Yoga practice is held between 2 weeks and 10 weeks, once a week, 5 times a week, 2 weeks and lasting approximately 25-45 minutes. In this study, the intervention will be implemented within 8 weeks. To the women who constitute the intervention group; After giving short-term self-care training in Menopause for 8 weeks, relaxation will be applied after the practice of Laughter yoga, which starts with breathing exercises, warm-up exercises, childlike games and has different exercises in each session. The research will be carried out in the Famagusta Municipality Development Academy, in a bright hall where women can take a U shape, everyone will be face to face, and will not be disturbed during the application.
  Interventions: Behavioral: Laughter Yoga
- Control Group (No Intervention): Routine care was given to the control group

INTERVENTIONS:
Behavioral: Laughter Yoga — Laughter yoga is a childlike practice where group members make eye contact with each other.
  It is a breath yoga practiced by imitating games and fake laughing. Brain the effects of real laughter on the body, as it cannot distinguish between fake and real laughter.
  showing positive effects. It consists of sessions lasting at least 20 minutes and an average of 45 minutes.
  Other Names: control
  Arms: Laughter Yoga Group

SUMMARY:
In order to evaluate the effects of laughter yoga on the quality of life, stress, cortisol, blood pressure levels and conscious self-care powers of menopausal women, it will be performed in two stages (the first stage is qualitative and the second stage is randomized controlled) on menopausal women in the TRNC Famagusta region.

DETAILED DESCRIPTION:
Menopause; It is defined as the cessation of menstrual bleeding and loss of ovarian function. The average age of entering menopause is known as 45-50. With the increase in life expectancy at birth in the world and in our country, women spend one third of their lives in the menopause period and are affected by the changes experienced during menopause for a longer period. For this reason, as life expectancy increases, it is important for women to take care of themselves and to take appropriate health care so that they can go through the menopause period well and improve their quality of life.

Due to the depletion of the estrogen hormone during menopause, many effects occur in women, many signs and symptoms are experienced, and daily life activities are significantly adversely affected. The type and severity of menopausal complaints in women are experienced differently depending on the decrease in estrogen levels. Commonly reported physical symptoms include emotional symptoms such as hot flashes, night sweats, and sleep problems. In addition, physical symptoms such as vaginal dryness, loss of libido, skin dryness, and joint pain are observed. Physical, psychological and social changes that negatively affect women's self-care and quality of life during menopause are quite complex, and the nursing approach in this period includes diagnosis, support and health education.

The changes that a woman experiences during menopause can negatively affect her mood and prevent her from taking care of herself. He may not want to do positive things about his health. Studies have shown that the menopausal period affects the quality of life self care; refers to behaviors performed to maintain health or maintain physical and emotional balance.

There are barriers and facilitators to self-care. These; experience and skills, motivation, cultural beliefs and values, self-confidence, habits, functional and cognitive abilities, support from others, and access to care. These factors are important for women to cope with the problems they face during menopause, to perform self-care and to increase their quality of life. Mental changes in this period vary according to the way a woman perceives menopause, the culture she lives in, and the personality traits of the woman. While this process is considered easy in some societies, it may be perceived as a source of stress in other societies. Although menopause is sometimes met with relaxation and peace, most women experience a sense of loss; feel that their self-esteem and self-esteem have decreased. Recognition and coping with the menopause period, which impairs women's ability to be happy, productive and harmonious, has an important place in women's healthy and unproblematic life during this period. In a study by Tümer and Kartal (2018) that included 152 women to determine the relationship between women's attitudes towards menopause and their menopausal complaints, it was found that women with menopause experienced the most psychological complaints.

It is thought that it may be important to highlight personal resources that can play a protective role in order to reduce the negative effects of the difficult conditions women are in during the menopause process. In this context, it is predicted that personal resources such as conscious self-care may have protective effects on women's well-being. During the transition to menopause, women are at higher risk of developing depression, stress, anxiety, and emotional distress. Relaxation techniques and exercise programs are used to reduce the level of stress experienced. Among them, the best stress-busting method is considered to be laughing. As a therapy, laughter has positive effects such as lowering blood pressure, reducing stress, increasing immunity, and reducing pain.

One of the alternative methods that can be used to improve psychological problems during menopause is Laughter yoga. Laughter therapy/yoga, Dr. It is a therapeutic approach that includes laughter and yoga exercises developed by Kataria in 1995 . The therapy provides laughter without any jokes, comedy or humor and supports the realization of a heartfelt laughter in individuals without the involvement of cognitive thinking. It is stated that laughter therapy has psychological and physiological effects on individuals. In studies examining the psychological effects; therapy was found to reduce anxiety, depression and stress levels. In a study conducted in the USA, the stress levels of nursing students after laughter therapy were examined and it was concluded that their stress levels decreased by decreasing from 112 points to 103. As seen in the study, it was found that laughter yoga was effective in the level of stress and decreased.

In a study examining the difference between optimism, self-esteem, and depression to confirm the effect of a laughter yoga program in menopausal women in Korea; Laughter yoga has been found to be effective in increasing optimism and self-esteem. It has been found that the depression of women in menopause decreases. It has been determined that laughter yoga practiced for 40 minutes twice a week (8 sessions) in a hospital reduces the depression scores of individuals and improves sleep quality. It has been reported that laughter increases the ability to control negative situations such as stress and turn negative emotions such as depression into positive ones. In a study conducted in Ankara, in the first year students of the Department of Nursing; It has been determined that the laughter yoga intervention is effective in reducing mental symptoms and salivary cortisol. When the literature is examined, studies focusing on the effect of laughter yoga on both stress reduction and quality of life have not been found.

Since the number of women living in the post-menopausal period increases with the increase in the life expectancy of women, it is thought that Laughter yoga, which does not pose health risks, may be effective in reducing the menopausal symptoms experienced by women, reducing stress and increasing their quality of life. In this study, it was thought to draw attention to the relationship and importance of these elements by revealing the effect of Laughter yoga practice on stress, menopausal symptoms, quality of life and self-care.

In this study, it is aimed to evaluate the effect of Laughter yoga on the quality of life, stress, cortisol, blood pressure levels and conscious self-care powers of menopausal women in the intervention group compared to the control group.

At the end of the study; between the control group and the intervention group; "Laughter Yoga and Self Care Training" applied to women in menopause

1. H01: There is no difference between the perceived stress scale mean scores. H11: There is a difference between the perceived stress scale mean scores
2. H02: There is no difference between the menopause-specific quality of life scale mean scores.

   H12: There is a difference between the menopause-specific quality of life scale mean scores. there is difference
3. H03: There is no difference between the mean scores of the self-care power scale.

   H13: There is a difference between the mean scores of the self-care power scale.
4. H04: There is no difference between the mean scores of the mindfulness-based self-care scale H14: There is a difference between the mean scores of the mindfulness-based self-care scale.
5. H05: No difference in salivary cortisol level H05: There is a difference in salivary cortisol level.
6. H06: No difference in blood pressure values H06: There is a difference in blood pressure values.

ELIGIBILITY:
Inclusion Criteria:

* Those who have been in menopause for the last five years
* At least 1 year past the last menstrual period
* Women between the ages of 45-60
* Willingness to participate in the research
* No communication barrier (cognitive affective)

Exclusion Criteria:

* Not knowing Turkish
* Having surgical menopause
* State their willingness to withdraw from the research voluntarily

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — menopausal women
Enrollment: 60 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-02-16 (Estimated); Study Completion 2024-02-16 (Estimated)

PRIMARY OUTCOMES:
The Effect of Laughter Yoga on Self-Care in Menopause | 8 WEEKS
  Conscious Awareness Based Self-Care Scale: The Conscious Awareness-Based Self-Care Scale developed by Cook-Cottone and Guyker (2018) is a multidimensional tool that examines self-care through the perceived involvement of individuals in the areas of physical, cognitive, emotional and social care and consists of 33 items. Conscious self-care is measured in six sub-dimensions: physical care, supportive relationships, mindfulness, self-compassion and purpose, conscious relaxation and supportive structure. The internal consistency coefficient was .89 for the general scale and .69, .86, .92, .83, .77, and .77 for the subscales, respectively. The Turkish validity and reliability study of the scale was carried out by Sünbül et al. (2018) and the internal consistency coefficient was .89 for the general scale and .72, .81, .81, .83, .66, and .80 for the subscales, respectively. E-mail permission has been obtained for the use of the scale.
The Effect of Laughter Yoga on Stress Level in Menopause | 8 WEEKS
  Perceived Stress Scale: The Perceived Stress Scale (PSS) was developed by Cohen, Kamarck, and Mermelstein in 1983. The scale consists of a total of 14 items and is designed to measure how stressful the individual perceives the situations in his life. Turkish validity and reliability studies of the scale were carried out by Eskin et al. in 2013. The items of the 14-item form preferred in this study are scored between 0-4. Scoring of the scale; Never (0), Almost never (1), Sometimes (2), Quite often (3), and Very often (4). The score of PSS-14 varies between 0-56; A high score means that the perception of stress is high. In scale; Items 4, 5, 6, 7, 9, 10 and 13 are reverse scored. The test-retest reliability coefficient of the scale was 0.87 and the cronbach alpha internal consistency coefficient was 0.84. E-mail permission was obtained for the use of the scale.
The Effect of Laughter Yoga on Quality of Life Scale Level in Menopause | 8 WEEKS
  Self-Care Strength Scale (PSAS): The scale used to measure an individual's self-care ability or self-care power was developed in English by Kearney and Fleicher (1979) with 43 items, and an abbreviated 35-item Turkish form was adapted by Nahcivan. The scale focused on individuals' self-assessment of their involvement in self-care actions. Each statement is scored from 0 to 4. In the Turkishized scale, 8 items (3, 6, 9, 13, 19, 22, 26 and 31) are evaluated as negative and the scoring is reversed. The maximum score is 140. The high score obtained from the scale indicates the high level of self-care or self-care ability and power of the individual. There is no cut off value. E-mail permission has been obtained for the use of the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Dilek Karaoğlan Gülevi, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR

REFERENCES:
- [Result] Treloar AE. Menstrual cyclicity and the pre-menopause. Maturitas. 1981 Dec;3(3-4):249-64. doi: 10.1016/0378-5122(81)90032-3. PMID 7334935
- [Result] Grindler NM, Santoro NF. Menopause and exercise. Menopause. 2015 Dec;22(12):1351-8. doi: 10.1097/GME.0000000000000536. PMID 26382311
- [Result] Sussman M, Trocio J, Best C, Mirkin S, Bushmakin AG, Yood R, Friedman M, Menzin J, Louie M. Prevalence of menopausal symptoms among mid-life women: findings from electronic medical records. BMC Womens Health. 2015 Aug 13;15:58. doi: 10.1186/s12905-015-0217-y. PMID 26271251
- [Result] Woods NF, Mitchell ES. Symptoms during the perimenopause: prevalence, severity, trajectory, and significance in women's lives. Am J Med. 2005 Dec 19;118 Suppl 12B:14-24. doi: 10.1016/j.amjmed.2005.09.031. PMID 16414323
- [Result] Thurston RC, Joffe H. Vasomotor symptoms and menopause: findings from the Study of Women's Health across the Nation. Obstet Gynecol Clin North Am. 2011 Sep;38(3):489-501. doi: 10.1016/j.ogc.2011.05.006. PMID 21961716
- [Result] Guerin E, Goldfield G, Prud'homme D. Trajectories of mood and stress and relationships with protective factors during the transition to menopause: results using latent class growth modeling in a Canadian cohort. Arch Womens Ment Health. 2017 Dec;20(6):733-745. doi: 10.1007/s00737-017-0755-4. Epub 2017 Jul 13. PMID 28707156